CLINICAL TRIAL: NCT06006156
Title: Long-term Dimensional Changes in Single Crowns Supported by Short (6 mm) Transmucosal Implants With Divergent or Convergent Neck Profiles in the Esthetic Zone. A Randomized Randomized Controlled Clinical Trial
Brief Title: Dimensional Changes in Single Crowns Supported by Short Transmucosal Implants With Diverging or Converging Neck Profiles in the Esthetic Zone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Collaborators: Universidad Nacional de Trujillo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNT_short implants
Record Dates: First submitted 2023-04-05; First posted 2023-08-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Maxilla; Partially edentulous; Dental implant; Implant supported prosthesis

STUDY DESIGN:
Intervention Model Description: The study is a split-mouth randomized controlled trial. One implant with a converging collar with micro threads or a diverging polished collar will be installed in each patient according to randomization in the esthetic region of the upper jaw ( between the second premolars ). It will be restored with individual crowns after three months of healing. Both implants will be placed with the rough margin of ~1 mm subcrestally.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment assignments will be sealed in opaque envelopes that will be opened during the surgery. The treatment assignment will be disclosed to the surgeon after the elevation of the alveolar mucosal flaps and prior to the preparation of the recipient sites.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dental implant with a convergent collar (Experimental): One implant with a converging collar with micro threads will be installed in each patient according to the site randomization in the esthetic region of the upper jaw (between the second premolars).
  Interventions: Procedure: Dental implants placement
- dental implant with a divergent collar (Active Comparator): One implant with a diverging polished collar will be installed in each patient according to the site randomization in the esthetic region of the upper jaw ( between the second premolars).
  Interventions: Procedure: Dental implants placement

INTERVENTIONS:
Procedure: Dental implants placement — surgery for placement of two one-piece trans gingival implants
  Other Names: implant supported prosthetic restoration

SUMMARY:
The goal of the present randomized clinical trial is to assess the long-term osseous and peri-implant soft tissue changes as well as the success rate of short implants (6 mm) with a converging collar with micro threads or a diverging polished collar placed in the esthetic zone of the maxilla on partially edentulous patients. The main questions it aims to answer are:

* what are the long-term bone and soft tissue changes around implants with a converging collar with micro threads compared to a diverging polished collar placed in the esthetic zone of the maxilla?
* What is the success rate of implants with a converging collar with micro threads compared to a diverging polished collar placed in the esthetic zone of the maxilla? Dental implants with a converging collar with micro threads or a diverging polished collar will be placed in the esthetic zone of the maxilla of the included participants and the measurements regarding the bone and soft tissue level will be compared.

DETAILED DESCRIPTION:
The objectives of the present randomized clinical trial are to evaluate the clinical and radiographic changes over time of hard and soft tissues around implants with a convergent or divergent collar. Twenty volunteer participants with two edentulous regions in the maxillary esthetic zone (from the right second premolar to the left second premolar) will be included in the study. Two implants will be randomly installed, one with a convergent collar and one with a divergent collar. After 3 months of healing, individual crowns will be installed. At each visit the following parameters will be evaluated: plaque index, probing depth, bleeding on probing, the recession of the mucosal margin, intraoral radiographs, likewise control CBCT, and impressions will be performed. The visit will take place at 6 and 12 months and then annually for a minimum of 3 years. Changes at the level of the marginal bone will be assessed overtime on the radiographs. Dimensional changes will be clinically evaluated during control evaluations and later through digital impressions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two edentulous areas in the esthetic region of the maxilla (from right to left from second premolar to premolar, preferably first premolars and incisors)
* Alveolar bone ≥ 8 mm in height and ≥ 5 mm in thickness assessed on CBCT.
* Age of ≥ 21 years.
* Need for an implant-supported prosthetic restoration.
* Be in good general health with no contraindications to oral surgical procedures.
* Not be pregnant.
* Patients who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* The presence of any uncontrolled systemic disease.
* History of past or ongoing chemotherapeutic or radiotherapeutic treatments.
* Heavy smokers (>10 cigarettes per day).
* Previous bone regeneration procedures in the area of interest

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
height of the periimplant bone tissues | baseline
  The height of the periimplant bone tissues will be evaluated in the intraoral radiographic images, cone beam tomography, and the three-dimensional images obtained from the digital prints
height of the periimplant bone tissues | 3 years follow up
  The height of the periimplant bone tissues will be evaluated in the intraoral radiographic images, cone beam tomography, and the three-dimensional images obtained from the digital prints
height of the periimplant soft tissues | Baseline
  The height of the periimplant soft tissues will be evaluated in the intraoral radiographic images, cone beam tomography, and the three-dimensional images obtained from the digital prints
height of the periimplant soft tissues | 3 years follow up
  The height of the periimplant soft tissues will be evaluated in the intraoral radiographic images, cone beam tomography, and the three-dimensional images obtained from the digital prints

SECONDARY OUTCOMES:
Plaque index | 1 year
  to score the plaque accumulation of plaque around implants will be used the Mombelli et al index
Plaque index | 3 year
  to score the plaque accumulation of plaque around implants will be used the Mombelli et al index
Bleeding on probing | 1 year
  During the probing, the bleeding on probing will be registered in the periodontal record.
Bleeding on probing | 3 year
  During the probing, the bleeding on probing will be registered in the periodontal record.
Probing depth | 1 year
  A calibrated probe will be used to measure the probing depth in all teeth annually.
Probing depth | 3 year
  A calibrated probe will be used to measure the probing depth in all teeth annually.
Implant success rate | 1 year
  The criteria to evaluate the success rate will be if there was no persistent and/or irreversible signs or symptoms such as pain, infection, neuropathies, or paresthesia, no peri-implant infection with suppuration, no mobility, and no continuous radiolucency around the implant.
Implant success rate | 3 years
  The criteria to evaluate the success rate will be if there was no persistent and/or irreversible signs or symptoms such as pain, infection, neuropathies, or paresthesia, no peri-implant infection with suppuration, no mobility, and no continuous radiolucency around the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Trujillo, Trujillo, La Libertad, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agustin-Panadero R, Martinez-Martinez N, Fernandez-Estevan L, Faus-Lopez J, Sola-Ruiz MF. Influence of Transmucosal Area Morphology on Peri-Implant Bone Loss in Tissue-Level Implants. Int J Oral Maxillofac Implants. 2019 July/August;(34):947-952. doi: 10.11607/jomi.7329. Epub 2019 Feb 15. PMID 30768662
- [Result] Altaib FH, Alqutaibi AY, Al-Fahd A, Eid S. Short dental implant as alternative to long implant with bone augmentation of the atrophic posterior ridge: a systematic review and meta-analysis of RCTs. Quintessence Int. 2019;50(8):636-650. doi: 10.3290/j.qi.a42948. PMID 31372602
- [Result] Bitaraf T, Keshtkar A, Rokn AR, Monzavi A, Geramy A, Hashemi K. Comparing short dental implant and standard dental implant in terms of marginal bone level changes: A systematic review and meta-analysis of randomized controlled trials. Clin Implant Dent Relat Res. 2019 Aug;21(4):796-812. doi: 10.1111/cid.12774. Epub 2019 May 1. PMID 31044538
- [Result] Buser D, Ingimarsson S, Dula K, Lussi A, Hirt HP, Belser UC. Long-term stability of osseointegrated implants in augmented bone: a 5-year prospective study in partially edentulous patients. Int J Periodontics Restorative Dent. 2002 Apr;22(2):109-17. PMID 12019706
- [Result] Caneva M, Lang NP, Calvo Guirado JL, Spriano S, Iezzi G, Botticelli D. Bone healing at bicortically installed implants with different surface configurations. An experimental study in rabbits. Clin Oral Implants Res. 2015 Mar;26(3):293-9. doi: 10.1111/clr.12475. Epub 2014 Sep 15. PMID 25220835
- [Result] Doyle AD, Wang FW, Matsumoto K, Yamada KM. One-dimensional topography underlies three-dimensional fibrillar cell migration. J Cell Biol. 2009 Feb 23;184(4):481-90. doi: 10.1083/jcb.200810041. Epub 2009 Feb 16. PMID 19221195
- [Result] Hermann JS, Jones AA, Bakaeen LG, Buser D, Schoolfield JD, Cochran DL. Influence of a machined collar on crestal bone changes around titanium implants: a histometric study in the canine mandible. J Periodontol. 2011 Sep;82(9):1329-38. doi: 10.1902/jop.2011.090728. Epub 2011 Apr 12. PMID 21486176
- [Result] Papaspyridakos P, De Souza A, Vazouras K, Gholami H, Pagni S, Weber HP. Survival rates of short dental implants (</=6 mm) compared with implants longer than 6 mm in posterior jaw areas: A meta-analysis. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:8-20. doi: 10.1111/clr.13289. PMID 30328206
- [Result] Ravida A, Majzoub J, Alassadi M, Saleh MH, Askar H, Wang HL. Impact of Implant Length on Survival of Rough-Surface Implants in Nonaugmented Posterior Areas: A Systematic Review and Meta-Regression Analysis. Int J Oral Maxillofac Implants. 2019 Nov/Dec;34(6):1359-1369. doi: 10.11607/jomi.7509. PMID 31711077
- [Result] Ravida A, Wang IC, Sammartino G, Barootchi S, Tattan M, Troiano G, Laino L, Marenzi G, Covani U, Wang HL. Prosthetic Rehabilitation of the Posterior Atrophic Maxilla, Short (</=6 mm) or Long (>/=10 mm) Dental Implants? A Systematic Review, Meta-analysis, and Trial Sequential Analysis: Naples Consensus Report Working Group A. Implant Dent. 2019 Dec;28(6):590-602. doi: 10.1097/ID.0000000000000919. PMID 31274666
- [Result] Rodriguez X, Navajas A, Vela X, Fortuno A, Jimenez J, Nevins M. Arrangement of Peri-implant Connective Tissue Fibers Around Platform-Switching Implants with Conical Abutments and Its Relationship to the Underlying Bone: A Human Histologic Study. Int J Periodontics Restorative Dent. 2016 Jul-Aug;36(4):533-40. doi: 10.11607/prd.2580. PMID 27333011
- [Result] Rossi F, Botticelli D, Cesaretti G, De Santis E, Storelli S, Lang NP. Use of short implants (6 mm) in a single-tooth replacement: a 5-year follow-up prospective randomized controlled multicenter clinical study. Clin Oral Implants Res. 2016 Apr;27(4):458-64. doi: 10.1111/clr.12564. Epub 2015 Feb 18. PMID 25692556
- [Result] Rossi F, Lang NP, Ricci E, Ferraioli L, Baldi N, Botticelli D. Long-term follow-up of single crowns supported by short, moderately rough implants-A prospective 10-year cohort study. Clin Oral Implants Res. 2018 Dec;29(12):1212-1219. doi: 10.1111/clr.13386. Epub 2018 Dec 6. PMID 30430655
- [Result] Rossi F, Lang NP, Ricci E, Ferraioli L, Marchetti C, Botticelli D. 6-mm-long implants loaded with fiber-reinforced composite resin-bonded fixed prostheses (FRCRBFDPs). A 5-year prospective study. Clin Oral Implants Res. 2017 Dec;28(12):1478-1483. doi: 10.1111/clr.13015. Epub 2017 Mar 28. PMID 28370406
- [Result] Storelli S, Abba A, Scanferla M, Botticelli D, Romeo E. 6 mm vs 10 mm-long implants in the rehabilitation of posterior jaws: A 10-year follow-up of a randomised controlled trial. Eur J Oral Implantol. 2018;11(3):283-292. PMID 30246182
- [Result] Szathvary I, Caneva M, Caneva M, Bressan E, Botticelli D, Meneghello R. A volumetric 3-D digital analysis of dimensional changes to the alveolar process at implants placed immediately into extraction sockets. J Oral Science Rehabilitation. 2015 Sep;1(1):62-9.
- [Result] Welander M, Abrahamsson I, Berglundh T. Subcrestal placement of two-part implants. Clin Oral Implants Res. 2009 Mar;20(3):226-31. doi: 10.1111/j.1600-0501.2008.01637.x. PMID 19397633

DOCUMENTS (1):
  • Study Protocol (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT06006156/Prot_000.pdf